CLINICAL TRIAL: NCT03341637
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Investigate the Immunogenicity and Safety of Subcutaneous Administration of a Tetravalent Dengue Vaccine Candidate in Healthy Adolescent Subjects in Non-Endemic Area(s) for Dengue
Brief Title: Immunogenicity and Safety of Tetravalent Dengue Vaccine (TDV) in Adolescents in Non-Endemic Area(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEN-315; U1111-1192-7827 (Other: World Health Organization); RNEC-2017-DEN-315 (Registry Identifier: Mexico); 2018-003980-77 (EudraCT Number)
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-07

CONDITIONS: Dengue
Keywords: Drug Therapy
MeSH Terms: conditions — Dengue | interventions — Dengue Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tetravalent Dengue Vaccine (TDV) (Experimental): TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose)
  Interventions: Biological: Tetravalent Dengue Vaccine (TDV)
- Placebo (Placebo Comparator): TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Tetravalent Dengue Vaccine (TDV) — TDV subcutaneous injection
  Arms: Tetravalent Dengue Vaccine (TDV)
Biological: Placebo — Normal Saline (0.9% NaCl) subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study was to describe the neutralizing antibody response against each dengue serotype at 1 month post second dose of TDV or placebo in dengue-naive adolescent participants.

DETAILED DESCRIPTION:
The vaccine tested in this study was tetravalent dengue vaccine (TDV). TDV was tested to assess the safety and immunogenicity in healthy adolescents in non-endemic area(s) for dengue.

The study enrolled 400 healthy participants. Participants were randomized in 3:1 ratio to receive:

* TDV 0.5 mL subcutaneous injection
* Placebo normal saline solution (0.9% NaCl) for injection.

In each trial group, participants received 2-dose schedule of TDV or placebo by subcutaneous injection on Days 1 (Month 0) and 90 (Month 3), but not all participants received both doses (8 subjects discontinued the trial before receiving the second dose).

This multi-center trial was conducted in Mexico. The overall time to participate in this study was 270 days. Participants had multiple visits to the clinic including a final visit at Day 270.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is aged 12 to 17 years, inclusive;
2. Is in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and the clinical judgment of the Investigator.
3. The participant/the participant's legally authorized representative (LAR) signs and dates a written, informed consent/assent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
4. Individuals who can comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. Has an elevated oral temperature (≥38°C or 100.4°F) within 3 days of the intended date of vaccination.
2. Known hypersensitivity or allergy to any of the vaccine components.
3. Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the Investigator, may interfere with the participant's ability to participate in the trial.
4. Has any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (e.g., Guillain-Barre syndrome).
5. History or any illness that, in the opinion of the Investigator, might interfere with the results of the trial or pose additional risk to the participant due to participation in the trial.
6. Has known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (M0) (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥ 2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (M0).
   3. Administration of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (M0) or planned administration during the trial.
   4. Receipt of immune-stimulants within 60 days prior to Day 1 (M0).
   5. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (M0).
   6. Human immunodeficiency virus (HIV) infection or HIV-related disease.
   7. Genetic immunodeficiency.
7. Has abnormalities of splenic or thymic function.
8. Has a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding.
9. Has any serious chronic or progressive disease according to judgment of the Investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
10. Has body mass index (BMI) greater than or equal to 35 kg/m^2 (= weight in kg/[height in square meters]).
11. Individuals participating in any clinical trial with another investigational product 30 days prior to Day 1 (M0) or intent to participate in another clinical trial at any time during the conduct of this trial.
12. Has received any other vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of trial vaccine administration.
13. Individuals involved in the trial conduct or their first degree relatives.
14. Has history of substance or alcohol abuse within the past 2 years.
15. Female participants who are pregnant or breastfeeding.
16. Females of childbearing potential who are sexually active, and who have not used any of the acceptable contraceptive methods for at least 2 months prior to Day 1 (M0).
17. Females of childbearing potential who are sexually active, and who refuse to use an acceptable contraceptive method up to 6 weeks after the last dose of trial vaccine. In addition, they must be advised not to donate ova during this period.
18. Any positive or indeterminate pregnancy test.
19. Previous and planned vaccination (during the trial conduct), against any flaviviruses including dengue, yellow fever (YF), Japanese encephalitis (JE) viruses or tick-borne encephalitis.
20. Previous participation in any clinical trial of a dengue or other flavivirus (eg, West Nile [WN] virus) candidate vaccine, except for participants who received placebo in those trials.
21. Participants with documented or suspected disease caused by a flavivirus such as dengue, Zika, YF, JE, WN fever, tick-borne encephalitis or Murray Valley encephalitis.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-01-26 (Actual); Study Completion 2019-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (5):
- Mexico (5):
  - Instituto Nacional de Pediatria (INP), Mexico City
  - Hospital Infantil de Mexico Federico Gomez, Mexico City
  - Biodextra, S.A. de C.V., Mexico City
  - Mexico Centre for Clinical Research, Mexico City
  - Centro de Atencion E Investigacion Medica (CAIMED) Mexico DF, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- [Derived] Biswal S, Mendez Galvan JF, Macias Parra M, Galan-Herrera JF, Carrascal Rodriguez MB, Rodriguez Bueno EP, Brose M, Rauscher M, LeFevre I, Wallace D, Borkowski A. Immunogenicity and safety of a tetravalent dengue vaccine in dengue-naive adolescents in Mexico City. Rev Panam Salud Publica. 2021 Jun 11;45:e67. doi: 10.26633/RPSP.2021.67. eCollection 2021. PMID 34131423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Mexico from 14-Dec-2017 to 26-Jan-2019.
Pre-assignment Details: Healthy volunteers were enrolled in a 3:1 ratio into 2 parallel study groups: 1 study group received 2 doses of Tetravalent Dengue vaccine (TDV) and another group received 2 doses of TDV matching placebo subcutaneously (SC).
Period: Overall Study
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Started | 100 | 300
Completed | 95 | 296
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Reason not Specified | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least 1 dose of trial vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV) | Total
Number analyzed (Participants) | 100 | 300 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.57) | 14.3 (1.69) | 14.3 (1.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 176 | 227
  Male | 49 | 124 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 100 | 300 | 400
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: If a participant had documented more than 1 race category on the case report form, the participant was only included under the multiracial category.
  Participants
    American Indian or Alaska Native | 55 | 148 | 203
    Multiracial | 45 | 152 | 197
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 100 | 300 | 400
Height [Mean (Standard Deviation); unit: cm] | 159.6 (8.94) | 159.0 (8.68) | 159.2 (8.74)
Weight [Mean (Standard Deviation); unit: kg] | 57.60 (14.045) | 56.84 (12.708) | 57.03 (13.041)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=Weight/Height.
  kg/m^2 | 22.42 (4.237) | 22.39 (4.266) | 22.40 (4.254)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Day 120
Description: GMTs of neutralizing antibodies were measured by microneutralization test 50% [MNT50] for each of the 4 Dengue Serotypes. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4. Seropositivity is defined as reciprocal neutralizing titer ≥10.
Time Frame: One month post second dose (Day 120)
Population: Per Protocol Set (PPS): all participants seronegative to all serotypes of dengue virus at baseline who received at least 1 dose of trial vaccine, who had a valid pre-dose (baseline) and at least 1 valid post-dose measurement for immunogenicity and no major protocol violations. Number analyzed: participants with data available at given time-point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 82 | 271
titer
  DENV-1: number analyzed (Participants) | 72 | 243
  DENV-1 | 5.3 [4.7 to 5.8] | 327.9 [281.7 to 381.8]
  DENV-2: number analyzed (Participants) | 72 | 243
  DENV-2 | 6.0 [5.2 to 7.0] | 1742.5 [1522.6 to 1994.3]
  DENV-3: number analyzed (Participants) | 72 | 243
  DENV-3 | 5.2 [4.8 to 5.6] | 119.5 [106.4 to 134.2]
  DENV-4: number analyzed (Participants) | 72 | 243
  DENV-4 | 5.1 [4.9 to 5.2] | 142.7 [126.4 to 161.0]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Day 270
Description: as for outcome 1
Time Frame: Six months post second dose (Day 270)
Population: PPS: all participants seronegative to all serotypes of dengue virus at baseline who received at least 1 dose of trial vaccine, who had a valid pre-dose (baseline) and at least 1 valid post-dose measurement for immunogenicity and no major protocol violations. Number analyzed: participants with data available at given time-point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 82 | 271
titer
  DENV-1: number analyzed (Participants) | 73 | 254
  DENV-1 | 5.4 [4.8 to 6.0] | 134.7 [114.5 to 158.5]
  DENV-2: number analyzed (Participants) | 73 | 254
  DENV-2 | 5.2 [4.8 to 5.5] | 740.9 [645.2 to 850.7]
  DENV-3: number analyzed (Participants) | 73 | 254
  DENV-3 | 5.3 [4.9 to 5.9] | 45.8 [40.7 to 51.5]
  DENV-4: number analyzed (Participants) | 73 | 254
  DENV-4 | 5.0 [NA to NA] — Data for 95% CI was not evaluable at this time point. | 37.5 [32.9 to 42.7]

3. Secondary Outcome: Seropositivity Rates for Each of the 4 Dengue Serotypes
Description: Seropositivity rate, defined as the percentage of participants seropositive, was derived from the titers of dengue-neutralizing antibodies. Seropositivity defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: One month and six months post second dose (Day 120 and Day 270)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 82 | 271
percentage of participants
  Day 120 (Month 4): DENV-1: number analyzed (Participants) | 72 | 243
  Day 120 (Month 4): DENV-1 | 1.4 [0.0 to 7.5] | 100.0 [98.5 to 100.0]
  Day 120 (Month 4): DENV-2: number analyzed (Participants) | 72 | 243
  Day 120 (Month 4): DENV-2 | 8.3 [3.1 to 17.3] | 100.0 [98.5 to 100.0]
  Day 120 (Month 4): DENV-3: number analyzed (Participants) | 72 | 243
  Day 120 (Month 4): DENV-3 | 1.4 [0.0 to 7.5] | 100.0 [98.5 to 100.0]
  Day 120 (Month 4): DENV-4: number analyzed (Participants) | 72 | 243
  Day 120 (Month 4): DENV-4 | 1.4 [0.0 to 7.5] | 99.6 [97.7 to 100.0]
  Day 270 (Month 9): DENV-1: number analyzed (Participants) | 73 | 254
  Day 270 (Month 9): DENV-1 | 2.7 [0.3 to 9.5] | 98.4 [96.0 to 99.6]
  Day 270 (Month 9): DENV-2: number analyzed (Participants) | 73 | 254
  Day 270 (Month 9): DENV-2 | 1.4 [0.0 to 7.4] | 99.6 [97.8 to 100.0]
  Day 270 (Month 9): DENV-3: number analyzed (Participants) | 73 | 254
  Day 270 (Month 9): DENV-3 | 2.7 [0.3 to 9.5] | 92.1 [88.1 to 95.1]
  Day 270 (Month 9): DENV-4: number analyzed (Participants) | 73 | 254
  Day 270 (Month 9): DENV-4 | 0 [0.0 to 4.9] | 89.4 [84.9 to 92.9]

4. Secondary Outcome: Seropositivity Rates for Multiple (2, 3 or 4) Dengue Serotypes
Description: Seropositivity rate, defined as the percentage of participants seropositive, was derived from the titers of dengue-neutralizing antibodies. Seropositivity was defined as a reciprocal neutralizing titer ≥10.
Time Frame: One month and six months post second dose (Day 120 and Day 270)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 82 | 271
percentage of participants
  Day 120 (Month 4): At Least Bivalent: number analyzed (Participants) | 72 | 243
  Day 120 (Month 4): At Least Bivalent | 1.4 [0.0 to 7.5] | 100.0 [98.5 to 100.0]
  Day 120 (Month 4): At Least Trivalent: number analyzed (Participants) | 72 | 243
  Day 120 (Month 4): At Least Trivalent | 1.4 [0.0 to 7.5] | 100.0 [98.5 to 100.0]
  Day 120 (Month 4): Tetravalent: number analyzed (Participants) | 72 | 243
  Day 120 (Month 4): Tetravalent | 1.4 [0.0 to 7.5] | 99.6 [97.7 to 100.0]
  Day 270 (Month 9): At Least Bivalent: number analyzed (Participants) | 73 | 254
  Day 270 (Month 9): At Least Bivalent | 0 [0.0 to 4.9] | 99.2 [97.2 to 99.9]
  Day 270 (Month 9): At Least Trivalent: number analyzed (Participants) | 73 | 254
  Day 270 (Month 9): At Least Trivalent | 0 [0.0 to 4.9] | 94.5 [90.9 to 97.0]
  Day 270 (Month 9): Tetravalent: number analyzed (Participants) | 73 | 254
  Day 270 (Month 9): Tetravalent | 0 [0.0 to 4.9] | 85.8 [80.9 to 89.9]

5. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary Recorded) Following Each Vaccination by Severity
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after vaccination and included pain (none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment and severe: prevents daily activity with or without treatment), redness (erythema) (<2.5 cm, mild: 2.5-5 cm, moderate: >5 to <=10 cm, severe: >10 cm) and swelling (edema/induration) (<2.5 cm, mild: 2.5-5 cm, moderate: >5 to <=10 cm, severe: >10 cm).
Time Frame: Within 7 days after each vaccination
Population: Safety Set included of all participants who received at least 1 dose of trial vaccine. Number analyzed is the number of participants with data available at the given timepoint. Only categories for which there was at least 1 participant are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 100 | 300
percentage of participants
  After First Vaccination, Any Solicited Local AEs: number analyzed (Participants) | 99 | 299
  After First Vaccination, Any Solicited Local AEs | 34.3 | 56.2
  After First Vaccination, Pain:Mild: number analyzed (Participants) | 99 | 299
  After First Vaccination, Pain:Mild | 26.3 | 44.8
  After First Vaccination, Pain:Moderate: number analyzed (Participants) | 99 | 299
  After First Vaccination, Pain:Moderate | 7.1 | 9.7
  After First Vaccination, Pain:Severe: number analyzed (Participants) | 99 | 299
  After First Vaccination, Pain:Severe | 1.0 | 0.7
  After First Vaccination, Erythema:Mild: number analyzed (Participants) | 99 | 299
  After First Vaccination, Erythema:Mild | 0 | 5.7
  After First Vaccination, Swelling:Mild: number analyzed (Participants) | 99 | 299
  After First Vaccination, Swelling:Mild | 0 | 4.3
  After Second Vaccination, Any Solicited Local AEs: number analyzed (Participants) | 94 | 295
  After Second Vaccination, Any Solicited Local AEs | 30.9 | 52.2
  After Second Vaccination, Pain:Mild: number analyzed (Participants) | 94 | 295
  After Second Vaccination, Pain:Mild | 24.5 | 35.6
  After Second Vaccination, Pain:Moderate: number analyzed (Participants) | 94 | 295
  After Second Vaccination, Pain:Moderate | 5.3 | 13.2
  After Second Vaccination, Pain:Severe: number analyzed (Participants) | 94 | 295
  After Second Vaccination, Pain:Severe | 1.1 | 3.1
  After Second Vaccination, Erythema:Mild: number analyzed (Participants) | 94 | 295
  After Second Vaccination, Erythema:Mild | 0 | 4.1
  After Second Vaccination, Swelling:Mild | 0 | 1.7
  After Second Vaccination, Swelling:Moderate | 0 | 0.3

6. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) (Diary Recorded) Following Each Vaccination by Severity
Description: Solicited systemic AEs were collected by participants using diary cards within 14 days after vaccination and included fever, headache, tiredness or weakness (asthenia), feeling of discomfort (malaise) and muscle pain (myalgia). Severity scales for headache were none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment and severe: prevents normal activity with or without treatment. Severity scales for others were none, mild: no interference with daily activity, moderate: interference with daily activity and severe: prevents daily activity. A systemic AE of fever (defined as ≥38°C or ≥100.4°F) was derived from a daily temperature reading recorded within 14 days after vaccination. Fever was excluded from the overall count as no severity grading was applied for it.
Time Frame: Within 14 days after each vaccination
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 100 | 300
percentage of participants
  After First Vaccination: Any Solicited Systemic AE: number analyzed (Participants) | 99 | 299
  After First Vaccination: Any Solicited Systemic AE | 58.6 | 66.6
  After First Vaccination: Headache-Mild: number analyzed (Participants) | 99 | 299
  After First Vaccination: Headache-Mild | 25.3 | 31.4
  After First Vaccination: Headache-Moderate: number analyzed (Participants) | 99 | 299
  After First Vaccination: Headache-Moderate | 18.2 | 10.4
  After First Vaccination: Headache-Severe: number analyzed (Participants) | 99 | 299
  After First Vaccination: Headache-Severe | 1.0 | 2.7
  After First Vaccination: Asthenia-Mild: number analyzed (Participants) | 99 | 299
  After First Vaccination: Asthenia-Mild | 20.2 | 24.7
  After First Vaccination: Asthenia-Moderate: number analyzed (Participants) | 99 | 299
  After First Vaccination: Asthenia-Moderate | 13.1 | 7.7
  After First Vaccination: Asthenia-Severe: number analyzed (Participants) | 99 | 299
  After First Vaccination: Asthenia-Severe | 2.0 | 2.3
  After First Vaccination: Malaise-Mild: number analyzed (Participants) | 99 | 299
  After First Vaccination: Malaise-Mild | 20.2 | 18.7
  After First Vaccination: Malaise-Moderate: number analyzed (Participants) | 99 | 299
  After First Vaccination: Malaise-Moderate | 11.1 | 7.7
  After First Vaccination: Malaise-Severe: number analyzed (Participants) | 99 | 299
  After First Vaccination: Malaise-Severe | 2.0 | 1.3
  After First Vaccination: Myalgia-Mild: number analyzed (Participants) | 99 | 299
  After First Vaccination: Myalgia-Mild | 26.3 | 36.1
  After First Vaccination: Myalgia-Moderate: number analyzed (Participants) | 99 | 299
  After First Vaccination: Myalgia-Moderate | 13.1 | 10.7
  After First Vaccination: Myalgia-Severe: number analyzed (Participants) | 99 | 299
  After First Vaccination: Myalgia-Severe | 1.0 | 1.0
  After First Vaccination:Fever-Any | 5.1 | 6.7
  After First Vaccination:Fever (38.0°C-<38.5°C): number analyzed (Participants) | 99 | 299
  After First Vaccination:Fever (38.0°C-<38.5°C) | 3.0 | 3.0
  After First Vaccination:Fever (38.5°C-<39.0°C): number analyzed (Participants) | 99 | 299
  After First Vaccination:Fever (38.5°C-<39.0°C) | 2.0 | 2.3
  After First Vaccination:Fever (39.0°C-<39.5°C): number analyzed (Participants) | 99 | 299
  After First Vaccination:Fever (39.0°C-<39.5°C) | 0.0 | 1.0
  After First Vaccination:Fever (39.5°C-<40.0°C): number analyzed (Participants) | 99 | 299
  After First Vaccination:Fever (39.5°C-<40.0°C) | 0.0 | 0.3
  After Second Vaccine: Any Solicited Systemic AEs: number analyzed (Participants) | 94 | 296
  After Second Vaccine: Any Solicited Systemic AEs | 45.7 | 49.3
  After Second Vaccination: Headache-Mild: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Headache-Mild | 20.2 | 24.3
  After Second Vaccination: Headache-Moderate: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Headache-Moderate | 6.4 | 8.4
  After Second Vaccination: Headache-Severe: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Headache-Severe | 3.2 | 2.7
  After Second Vaccination: Asthenia-Mild: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Asthenia-Mild | 22.3 | 19.9
  After Second Vaccination: Asthenia-Moderate: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Asthenia-Moderate | 4.3 | 6.8
  After Second Vaccination: Asthenia-Severe: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Asthenia-Severe | 1.1 | 1.4
  After Second Vaccination: Malaise-Mild: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Malaise-Mild | 12.8 | 16.2
  After Second Vaccination: Malaise-Moderate: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Malaise-Moderate | 6.4 | 5.1
  After Second Vaccination: Malaise-Severe: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Malaise-Severe | 4.3 | 2.4
  After Second Vaccination: Myalgia-Mild: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Myalgia-Mild | 21.3 | 25.7
  After Second Vaccination: Myalgia-Moderate: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Myalgia-Moderate | 8.5 | 6.8
  After Second Vaccination: Myalgia-Severe: number analyzed (Participants) | 94 | 296
  After Second Vaccination: Myalgia-Severe | 1.1 | 2.4
  After Second Vaccination:Fever-Any | 3.2 | 6.8
  After Second Vaccination:Fever (38.0°C-<38.5°C): number analyzed (Participants) | 94 | 296
  After Second Vaccination:Fever (38.0°C-<38.5°C) | 1.1 | 3.7
  After Second Vaccination:Fever (38.5°C-<39.0°C): number analyzed (Participants) | 94 | 296
  After Second Vaccination:Fever (38.5°C-<39.0°C) | 1.1 | 2.0
  After Second Vaccination:Fever (39.0°C-<39.5°C) | 1.1 | 0.7
  After Second Vaccination:Fever (39.5°C-<40.0°C) | 0.0 | 0.3

7. Secondary Outcome: Percentage of Participants With Any Unsolicited Adverse Events (AEs) Following Each Vaccination
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: Within 28 days after each vaccination
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 100 | 300
percentage of participants
  After First Vaccination | 25.0 | 30.0
  After Second Vaccination: number analyzed (Participants) | 95 | 297
  After Second Vaccination | 17.9 | 23.2

8. Secondary Outcome: Percentage of Participants With Medically Attended AEs (MAAEs) Throughout the Study
Description: MAAEs were defined as AEs leading to a medical visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria.
Time Frame: From first vaccination (Day 1) through end of study (Day 270)
Population: Safety Set included of all participants who received at least 1 dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 100 | 300
percentage of participants | 38.0 | 47.3

9. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Throughout the Study
Description: An SAE was defined as any untoward medical occurrence or effect that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: From first vaccination (Day 1) through end of study (Day 270)
Population: Safety Set included of all participants who received at least 1 dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 100 | 300
percentage of participants | 2.0 | 0.3

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: Within 28 days after Vaccination; MAAEs and SAEs: From first vaccination (Day 1) through end of study (Day 270)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Tetravalent Dengue Vaccine (TDV)
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/300
Serious Adverse Events (participants affected / at risk) | 2/100 | 1/300
Other Adverse Events (participants affected / at risk) | 38/100 | 112/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | Tetravalent Dengue Vaccine (TDV) (N=300)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | Tetravalent Dengue Vaccine (TDV) (N=300)
Viral upper respiratory tract infection (Infections and infestations) | 14 | 43
Nasopharyngitis (Infections and infestations) | 6 | 24
Viral pharyngitis (Infections and infestations) | 7 | 15
Pharyngitis (Infections and infestations) | 4 | 10
Pharyngitis bacterial (Infections and infestations) | 2 | 9
Gastroenteritis (Infections and infestations) | 2 | 8
Gastritis (Gastrointestinal disorders) | 3 | 7
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 9
Syncope (Nervous system disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-03-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT03341637/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03341637/SAP_001.pdf